CLINICAL TRIAL: NCT02043834
Title: Promoting Virtual Reality-based Exercise to Prevent Falls in Older Adults: Pilot Study
Brief Title: Virtual Reality-based Exercise in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARPF-123
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Distorted; Balance; Motor Deficit
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance Training (Experimental): Balance training will be conducted individually two times per week for 4 weeks. Each training session will include virtual reality tasks such as "ankle reaching" and "obstacle crossing" using a virtual obstacle shown on a computer screen. Each session will last 30 - 45 minutes.
  Interventions: Other: Balance Training
- Control (No Intervention): The control group will keep their normal activity without receiving any intervention.

INTERVENTIONS:
Other: Balance Training — Balance training will be conducted individually two times per week for 4 weeks. Each training session will include virtual reality tasks such as "ankle reaching" and "obstacle crossing" using a virtual obstacle shown on a computer screen. Each session will last 30 - 45 minutes.
  Arms: Balance Training

SUMMARY:
The aim of the present study is to evaluate an innovative virtual reality-based balance training intervention for improving clinically relevant motor performances (balance and gait) in older adults.

We hypothesize that the virtual reality-based balance training intervention will improve balance and gait performances in older adults compared to a control group receiving usual care only.

ELIGIBILITY:
Inclusion Criteria:

* ability to ambulate without assistance
* willingness to provide informed consent

Exclusion Criteria:

* severe neurologic, cardiovascular, metabolic, or psychiatric disorders
* severe visual impairment
* cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Postural Balance | after 4 weeks
  Postural Balance during quiet standing for 30 seconds will be assessed using validated wearable sensor technologies (BalanSens™)

SECONDARY OUTCOMES:
Gait performance | 4 weeks
  Gait performance will be measured using validated wearable sensor technology (LEGSys™)
Cognitive status | 4 weeks
  Changes in cognitive status will be measured by the Trail Making Test and the Category Fluency Test
Quality of life | 4 weeks
Functional performance | 4 weeks
  Functional performance will be assessed using the Timed Up and Go Test and the Alternate Step Test

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Najafi, PhD, Principal Investigator — interdisciplinary Consortium on Advanced Motion Performance (iCAMP), Department of Surgery, College of Medicine, University of Arizona; Michael Schwenk, PhD, Principal Investigator — interdisciplinary Consortium on Advanced Motion Performance (iCAMP), Department of Surgery, College of Medicine, University of Arizon
Locations (1):
- Villa Hermosa - Senior Living Tucson, Tucson, Arizona, United States

REFERENCES:
- [Derived] Schwenk M, Grewal GS, Honarvar B, Schwenk S, Mohler J, Khalsa DS, Najafi B. Interactive balance training integrating sensor-based visual feedback of movement performance: a pilot study in older adults. J Neuroeng Rehabil. 2014 Dec 13;11:164. doi: 10.1186/1743-0003-11-164. PMID 25496052